CLINICAL TRIAL: NCT02884154
Title: Feasibility and Yield of a New 20 G ProCore Needle With Coiled Sheath in the Gastrointestinal Subepithelial Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Gwang Ha Kim, Principal Investigator, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K_EUS_Study_1
Record Dates: First submitted 2016-08-21; First posted 2016-08-30 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal Tract; Gastrointestinal Stromal Tumor
Keywords: Endoscopic ultrasonography; Biopsy; Gastrointestinal tract; Subepithelial tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

ARMS (1):
- Arm who will undergo EUS-FNB (Other)
  Interventions: Device: Echotip ProCoreⓇ HD Ultrasound Biopsy Needle

INTERVENTIONS:
Device: Echotip ProCoreⓇ HD Ultrasound Biopsy Needle

SUMMARY:
The exact incidence of subepithelial tumors (SETs) in the gastrointestinal (GI) tract is unknown, but the prevalence of gastric SETs detected during routine esophagogastroduodenoscopy is 0.36%. GI SETs may include leiomyoma, GI stromal tumor (GIST), schwannoma, lipoma, cyst, or ectopic pancreas. Surgical resection is the principal diagnostic and therapeutic method for SETs, especially for large and symptomatic ones. Preoperative pathological diagnosis of SETs may facilitate clinical decision making, but conventional endoscopic forceps biopsy does not yield adequate amounts of subepithelial tissue for definitive diagnosis.

Although endoscopic ultrasonography (EUS) is the best imaging modality for the evaluation of SETs, it cannot substitute histopathological diagnosis. EUS-guided fine-needle aspiration (EUS-FNA) may provide adequate amounts of tissue for the diagnosis of SETs, but it does not always afford adequate samples for immunohistochemical analysis because of the often small number of cells obtained by aspiration. Since some SETs, especially GI mesenchymal tumors such as GIST or schwannoma, have varied morphologic appearances, and diagnosis using a small biopsy is not straightforward, immunohistochemical analysis is strongly advisable, if not essential. EUS-guided Trucut biopsy (EUS-TNB) may overcome the limitations of EUS-FNA in procuring sufficient core tissue specimens. Although EUS-TNB is more accurate than EUS-FNA for diagnosing GI mesenchymal tumors, the rigidity of its 19-gauge (G) caliber and the mechanical friction of the firing mechanism produced by the torqued echoendoscope limit its use for SETs located in the gastric antrum and duodenum. Therefore, a needle facilitating adequate histological core sampling with easy maneuverability needs to be established. A 19G EUS-guided fine-needle biopsy (EUS-FNB) device with ProCore reverse-bevel technology was recently introduced. A multicenter study revealed that histological samples could be successfully obtained using this needle in most patients having GI SETs, with a diagnostic accuracy of >80%.10 However, because of technical difficulties with this needle in the gastric antrum and duodenum, the same FNB device was recently developed in a 20 G platform with coiled sheath. This prospective, multicenter study aimed to evaluate feasibility, yield, and diagnostic accuracy of a newly developed 20 G ProCore needle with coiled sheath in patients with GI SETs.

DETAILED DESCRIPTION:
Patients and Methods

Patients with newly diagnosed GI SETs will be prospectively enrolled at 8 university hospitals in Korea between May and December 2016, if they met the following criteria: having a hypoechoic mass in the submucosal and/or proper muscle layers on the basis of EUS and tumor >2 cm in size. Exclusion criteria are: SETs were not located in the submucosal and/or proper muscle layers on EUS; EUS revealed the characteristic findings of lipoma, cyst, vessel or extraluminal lesions; the platelet count was <50,000/mm3 and prothrombin time was <50%; or the patient did not provide consent to undergo the study. This study is approved by the Institutional Review Board of each hospital and conducted in accordance with the Declaration of Helsinki and its amendments and the Good Clinical Practice guidelines. All enrolled patients provide written informed consents to participate in the study.

Technique for EUS-FNB

All procedures are performed by using a linear array echoendoscope (Olympus UCT-140, UCT-240; Olympus, Tokyo, Japan or PentaxEG-3870UTK; Pentax, Tokyo, Japan) with the patients placed in the left lateral decubitus position under conscious sedation.

Before the study commenced, all participating endosonographers discuss the procedural steps in detail. Technical details of the standard tissue-acquisition protocol are as follows. After the target lesion is endosonographically visualized and the region scanned for SETs using color or pulsed Doppler, FNB is performed at the esophagus, stomach, duodenum or rectum, depending on the lesion location. The needle is advanced into the target tissue under endosonographic guidance.

After penetrating the lesion, the endosonographer moves the needle to-and-fro for more than 10 to 15 times within the lesion while an assistant simultaneously pulled out the stylet slowly and continuously over 20 s to achieve minimal negative pressure within the needle (slow-pull technique). Finally, the needle is withdrawn from the lesion. At least three needle passes are performed using the designated needle, and if a diagnostic or technical failure is encountered, the patient is switched to the alternative needle according to the judgment of the endosonographers.

Preparation for histological analysis

Because pathologists are absent during endoscopy, FNB samples are recovered and stored for subsequent processing by the endosonographers. The specimens are then expressed onto slides by using a stylet or by flushing with air into the needle assembly, to harvest the core samples from the needle. The endosonographers then carefully inspect the material on the slides for the presence of tissue cores defined as whitish pieces of tissue with apparent bulk, which are measured and then lifted off the slides and placed into a formalin bottle. The core samples are macroscopically assessed as a definite tissue core; suspicious tissue core mixed with blood clots; or only blood or scarce sample without any tissue core. The former two sample types are considered macroscopically optimal core samples.

If tissue cores are obtained, they are fixed in formalin and stained in hematoxylin and eosin for evaluation by pathologists. Samples with tissue cores are graded as optimal or suboptimal: optimal, if the material allows satisfactory assessment of histologic architecture and immunohistochemical evaluation, such as c-kit, CD34, S-100, or smooth muscle actin, if indicated, and suboptimal, if the histological core is inadequate for the abovementioned assessments. Because the morphological characteristics of mesenchymal tumors are nonspecific, a positive diagnosis by EUS-FNB is only considered true positive when immunohistochemical analysis is conclusive. Conventional cytological analysis is additionally performed in most cases or if a core sample is unavailable. Cytological material is sent to the cytologists as a fixed or an air-dried slide. The gold standard is the histopathological assessment of the resected specimens for patients who underwent endoscopic resection or surgery, and the assessment of the FNB samples for those who did not.

Outcome parameters

The primary outcome parameter is diagnostic sufficiency. Diagnostic sufficiency is defined as the proportion of patients in whom the histopathological diagnosis could be established within three needle passes. The percentage of cases in which the pathologist classified the quality of the sample as optimal for histological evaluation is also evaluated. The secondary outcome measures are rates of diagnostic failure, technical failure, and complications. Diagnostic failure is defined as failure to obtain sufficient core samples even after three passes, and technical failure is defined as malfunction of the needle before three needle passes. Complications are defined as any deviation from the clinical course after EUS-guided sampling, as observed by the endosonographers or recovery suite nurses, or as reported by patients. Excessive bleeding at the site of puncture, perforation, hypotension, and need for reversal medication are documented.

ELIGIBILITY:
Inclusion Criteria:

* Having a hypoechoic mass in the submucosal and/or proper muscle layers on the basis of EUS and tumor >2 cm in size

Exclusion Criteria:

* SETs were not located in the submucosal and/or proper muscle layers on EUS
* EUS revealed the characteristic findings of lipoma, cyst, vessel or extraluminal lesions; the platelet count was <50,000/mm3 and prothrombin time was <50%
* The patient did not provide consent to undergo the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
diagnostic sufficiency | up to 2 weeks
  Diagnostic sufficiency is defined as the proportion of patients in whom the histopathological diagnosis could be established within three needle passes.

SECONDARY OUTCOMES:
diagnostic failure rate | up to 2 weeks
technical failure rate | up to 1 day
complications | up to 4 weeks

REFERENCES:
- [Derived] Kim DH, Kim GH, Cho CM, Park CH, Na SY, Kim TH, Cho YK, Kim JH, Seo DW; Korean EUS Study Group. Feasibility of a 20-gauge ProCore needle in EUS-guided subepithelial tumor sampling: a prospective multicenter study. BMC Gastroenterol. 2018 Oct 19;18(1):151. doi: 10.1186/s12876-018-0880-1. PMID 30340469